CLINICAL TRIAL: NCT00325260
Title: A Randomized, Endpoint-Blind, Parallel Group Study to Demonstrate the Non-Inferiority of the Subunit Influenza Vaccine Influvac® to the Subunit Influenza Vaccine Agrippal® in Healthy Children, Adults and Elderly in China.
Brief Title: Non-Inferiority Study Comparing the Subunit Vaccines Influvac and Agrippal in China
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: S201.3.121
Record Dates: First submitted 2006-05-11; First posted 2006-05-12 (Estimated); Last update posted 2006-11-01 (Estimated); Status verified 2006-10

CONDITIONS: Healthy
Keywords: influenza; non-inferiority; Influvac; Agrippal; healthy subjects
MeSH Terms: conditions — Influenza, Human | interventions — influvac

INTERVENTIONS:
Biological: Influvac; subunit influenza vaccine

SUMMARY:
In the study Influvac will be compared to Agrippal, another subunit influenza vaccine that is already on the market in China. The main objective of the study is to show that both vaccines are comparable with regard to efficacy. In addition, safety and efficacy data with Influvac will be assessed in the Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* signed and dated informed consent
* being healthy
* mental health enough to understand the study, the informed consent form and the questionnaire

Exclusion Criteria:

* known to be allergic to constituents of the vaccine
* having an autoimmune disorder, taking immunomodulating drugs or having immune disfunction secondary to HIV
* having had a documented serious adverse reaction to previous influenza vaccination
* having had documented influenza infection or vaccination in the six months prior to the start of the study
* having received any other vaccines, immunoglobulins or investigational drugs in the month prior to the start of the study

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 900
Dates: Start 2006-03

PRIMARY OUTCOMES:
HI titers 4 weeks after vaccination (efficacy) and safety and tolerability

SECONDARY OUTCOMES:
HI derived parameters: seroprotection, seroconversion and mean fold increase 4 weeks after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (1):
- Site 1, Nanjing, China